CLINICAL TRIAL: NCT04850365
Title: Comparison Between Abdominal Sacral Hysteropexy and Vaginal Sacrospinous Hysteropexy for Management of Women With Apical Uterine Descent : a Randomized Clinical Trial
Brief Title: Abdominal Sacral Hysteropexy Versus Vaginal Sacrospinous Hysteropexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Mostafa, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abdovagpexy
Record Dates: First submitted 2021-03-26; First posted 2021-04-20 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal sacral hysteropexy (Other): The approach involves suspending the cervix to the anterior longitudinal ligament on the sacrum using permanent sutures or polypropylene mesh.
  Interventions: Procedure: Hysteropexy
- Vaginal sacrospinous hysteropexy (Other): This transvaginal extraperitoneal technique involves suspending the sacrospinous ligament to the cervix using either a dissolvable or permanent suture. The suspension is performed in a unilateral fashion.
  The outcomes will be obtained as follow;
  Interventions: Procedure: Hysteropexy

INTERVENTIONS:
Procedure: Hysteropexy — Abdominal Sacral cervicopexy:
  The approach involves suspending the cervix to the anterior longitudinal ligament on the sacrum using permanent sutures or polypropylene mesh.
  Vaginal Sacrospinous cervicopexy:
  This transvaginal extraperitoneal technique involves suspending the sacrospinous ligament to the cervix using either a dissolvable or permanent suture. The suspension is performed in a unilateral fashion.

SUMMARY:
The aim of the current study is to compare abdominal sacral cervicopexy with vaginal sacrospinous cervicopexy in women with apical prolapse in terms of operative time, procedures safety and efficacy.

DETAILED DESCRIPTION:
According to Cochrane group trials , abdominal approaches centered on sacral colpopexy is associated with lower risk of awareness of prolapse, repeat surgery for prolapse and dyspareunia than a variety of vaginal interventions. However, these trials weren't statistically significant and have focused on the effects in terms of anatomy and lacked the effect on functional outcomes, the quality of life, perioperative complications and the operative duration.

In this study, We hypothesize that prolonged operative duration will be associated with a greater risk of developing complications and so may guide us to a minimally invasive approach with better functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:

  1. Symptomatic apical descent stage II or more.
  2. Eligible for both surgical procedures
  3. No uterine or cervical pathology.
  4. Able to consent to participate in the trial.

Exclusion Criteria:

1. Women with contraindication to any surgical procedures.
2. Women with previous apical prolapse surgery.
3. One of the two surgical approaches is not feasible.
4. Women with concomitant surgical procedures apart from correction of the prolapse.
5. Women who prefer to have hysterectomy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Operative time | intraoperative
  Operative time will be recorded starting from skin incision.

SECONDARY OUTCOMES:
a_clinical effectiveness assessed by the pelvic organ prolapse quantification system (POP_Q). | From 6 months to 1 year follow up
  The patients will be followed for recurrence of the symptoms and the degree of descent.
b_Number of participants with treatment_related adverse events as assessed by CTCAE v4.0 | From 6 months to 1 year follow up
  It will be used to assess the safety and tolerability to the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Ragab Mady, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt